CLINICAL TRIAL: NCT06484530
Title: Gene-guided N-acetyl Cysteine for Prophylaxis of Anti-tuberculous Drug- Induced Hepatitis: A Randomized Controlled Trial
Brief Title: Gene-guided N-acetyl Cysteine for Prophylaxis of Anti-tuberculous Drug- Induced Hepatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Si 708/2023
Record Dates: First submitted 2024-04-03; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis (TB); Isoniazid Toxicity; Rifampicin Toxicity; Pyrazinamide Adverse Reaction; Ethambutol Toxicity; NAT2 Slow Acetylator Status; NAT2 Rapid Acetylator Status; NAT2 Polymorphism; N-Acetylcysteine
Keywords: Tuberculosis (TB); Isoniazid Toxicity; Rifampicin Toxicity; Pyrazinamide Adverse Reaction; Ethambutol Toxicity; NAT2 Slow Acetylator Status; NAT2 Rapid Acetylator Status; NAT2 Polymorphism; N-Acetylcysteine
MeSH Terms: conditions — Tuberculosis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Patients with tuberculosis who meet the research criteria will be randomly assigned into 2 groups using a block of four method with a 1:1 ratio. Patients in group 1 will undergo NAT2 gene testing before starting anti-tuberculosis medication. If the NAT2 gene phenotype is identified as slow acetylator, the patient will receive NAC medication at a dose of 600 mg twice daily for 8 weeks in addition to anti-tuberculosis medication. If the NAT2 gene phenotype is identified as rapid or intermediate acetylator, the patient will receive only anti-tuberculosis medication. Patients in group 2 will receive standard anti-tuberculosis medication without NAT2 gene testing.All patients will undergo blood tests to monitor liver function, kidney function, and blood count at 2, 8 weeks, and 6 months after starting medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAT2 gene testing group (Experimental): Tuberculosis patients will undergo NAT2 gene testing before starting anti-tuberculosis medication. If the NAT2 gene phenotype is identified as slow acetylator, the patient will receive NAC medication at a dose of 600 mg twice daily for 8 weeks in addition to anti-tuberculosis medication. If the NAT2 gene phenotype is identified as rapid or intermediate acetylator, the patient will receive only anti-tuberculosis medication.
  Interventions: Drug: N acetyl cysteine
- Non NAT2 gene testing (No Intervention): Tuberculosis patients will receive standard anti-tuberculosis medication without NAT2 gene testing.

INTERVENTIONS:
Drug: N acetyl cysteine — 1,200 mg/day for 8 weeks in NAT2 gene testing group and NAT2 gene phenotype is identified as slow acetylator.
  Other Names: Standard anti TB drug regimen
  Arms: NAT2 gene testing group

SUMMARY:
Tuberculosis (TB) remains a significant public health concern in Thailand and globally, especially in tropical regions, with pulmonary TB being predominant. Besides affecting the lungs, TB can also impact extrapulmonary organs. Standard TB treatment involves a combination of drugs administered for at least 6 months, but it can cause adverse effects such as hepatitis. Hepatotoxicity, occurring in 20-60% of patients, is commonly linked to isoniazid, rifampicin, and pyrazinamide. Slow acetylators of the NAT2 gene are particularly susceptible. Previous research suggests N-acetylcysteine (NAC) may mitigate hepatotoxicity, especially among slow acetylators. A recent study by Kittichai Samaithongcharoen and team showed that NAC reduced hepatotoxicity incidence significantly among slow acetylators. This underscores the potential of NAC in preventing drug-induced hepatotoxicity in TB treatment, warranting further investigation against standard treatment protocols.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a significant public health problem in Thailand and globally, especially in hot climates. TB infection is commonly found in the lungs, but it can also affect other important organs such as lymph nodes, pleura, abdomen, musculoskeletal system, urinary tract, and nervous system. The current standard treatment regimen for TB consists of a combination of drugs (isoniazid, rifampicin, pyrazinamide, and ethambutol), used for new TB patients who have not been treated before or have received less than 1 month of treatment. A major challenge in TB treatment is that patients must take multiple drugs continuously for at least 6 months, with common side effects including skin rash, dizziness, hepatitis, nausea, vomiting, and abdominal pain, often occurring within the first 2 months of treatment. Hepatotoxicity from anti-TB drugs is a common side effect, occurring in 20-60% of patients, mostly within the first 2 weeks to 2 months of starting treatment. Isoniazid, rifampicin, and pyrazinamide are the drugs most commonly associated with hepatotoxicity, typically causing hepatocellular injury of varying severity. NAT2 slow acetylator phenotype individuals are at higher risk. Studies in Thailand have found a high prevalence (25-30%) of NAT2 slow acetylators among Thai people. Preventing hepatotoxicity from anti-TB drugs is crucial, especially for high-risk patients, although clear guidelines are lacking. Previous studies have shown that administering N-acetylcysteine (NAC), an antioxidant, can reduce hepatotoxicity, particularly in slow acetylators. A recent controlled study by Kittichai Samaithongcharoen and colleagues demonstrated the significant efficacy of NAC in preventing hepatotoxicity in slow acetylators receiving standard TB treatment, with no cases of hepatotoxicity compared to a 50% incidence in the control group. Further research is needed to explore the effectiveness of NAC administration for preventing hepatotoxicity from anti-TB drugs, based on NAT2 genotype testing, compared to current standard TB treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 80 years old.
* Newly diagnosed tuberculosis patients (both pulmonary and extrapulmonary).
* Received standard anti-tuberculosis medication according to standard regimens (2HRZE/4HR, 2HRE/7HR).
* Willing to participate in the research

Exclusion Criteria:

* Infected with HIV.
* Severe liver dysfunction classified as Child-Pugh B or C.
* Chronic untreated liver diseases such as hepatitis B or C, alcoholic liver disease.
* Abnormal liver function tests including AST > 1.5 times the upper limit of normal (48 U/L), ALT > 1.5 times the upper limit of normal (55 U/L), ALP > upper limit of normal (110 U/L), Total bilirubin > upper limit of normal (1.2 mg/dL).
* Diagnosed with cancer.
* History of allergy to N-acetylcysteine (NAC).
* Pregnant or breastfeeding.
* Severe comorbidities such as CKD stage 4-5, chronic heart failure, severe pulmonary diseases (COPD, bronchiectasis).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hepatitis at 8 weeks | 8 weeks
  To study the efficacy of administering N-acetylcysteine (NAC) to prevent drug-induced hepatitis at 8 weeks from anti-tuberculosis medication using gene-guided therapy compared to conventional therapy.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels or Total bilirubin(TB) more than 2.5 milligrams per decilitre (mg/dL)

SECONDARY OUTCOMES:
Prevalence of hepatitis at 2 weeks | 2 weeks
  To study the efficacy of administering N-acetylcysteine (NAC) to prevent drug-induced hepatitis at 2 weeks from anti-tuberculosis medication using gene-guided therapy compared to conventional therapy.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels or Total bilirubin(TB) more than 2.5 milligrams per decilitre (mg/dL)

OTHER OUTCOMES:
Prevalence of hepatitis at 24 weeks | 24 weeks
  To study the efficacy of administering N-acetylcysteine (NAC) to prevent drug-induced hepatitis at 24 weeks from anti-tuberculosis medication using gene-guided therapy compared to conventional therapy.
  Significant hepatitis was defined as elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 5 times of baseline levels or Total bilirubin(TB) more than 2.5 milligrams per decilitre (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Supot Nimanong, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Background] Palwatwichai A. Tuberculosis in Thailand. Respirology. 2001 Mar;6(1):65-70. doi: 10.1046/j.1440-1843.2001.00299.x. PMID 11264766
- [Background] Treatment of Tuberculosis: Guidelines. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138748/ PMID 23741786
- [Background] Wiwatworapan T, Anantasetagoon T. Extra-pulmonary tuberculosis at a regional hospital in Thailand. Southeast Asian J Trop Med Public Health. 2008 May;39(3):521-5. PMID 18564694
- [Background] Bouazzi OE, Hammi S, Bourkadi JE, Tebaa A, Tanani DS, Soulaymani-Bencheikh R, Badrane N, Bengueddour R. First line anti-tuberculosis induced hepatotoxicity: incidence and risk factors. Pan Afr Med J. 2016 Nov 16;25:167. doi: 10.11604/pamj.2016.25.167.10060. eCollection 2016. PMID 28292129
- [Background] Anand AC, Seth AK, Paul M, Puri P. Risk Factors of Hepatotoxicity During Anti-tuberculosis Treatment. Med J Armed Forces India. 2006 Jan;62(1):45-9. doi: 10.1016/S0377-1237(06)80155-3. Epub 2011 Jul 21. PMID 27407844
- [Background] Gaude GS, Chaudhury A, Hattiholi J. Drug-induced hepatitis and the risk factors for liver injury in pulmonary tuberculosis patients. J Family Med Prim Care. 2015 Apr-Jun;4(2):238-43. doi: 10.4103/2249-4863.154661. PMID 25949974
- [Background] Ramappa V, Aithal GP. Hepatotoxicity Related to Anti-tuberculosis Drugs: Mechanisms and Management. J Clin Exp Hepatol. 2013 Mar;3(1):37-49. doi: 10.1016/j.jceh.2012.12.001. Epub 2012 Dec 20. PMID 25755470
- [Background] Ostapowicz G, Fontana RJ, Schiodt FV, Larson A, Davern TJ, Han SH, McCashland TM, Shakil AO, Hay JE, Hynan L, Crippin JS, Blei AT, Samuel G, Reisch J, Lee WM; U.S. Acute Liver Failure Study Group. Results of a prospective study of acute liver failure at 17 tertiary care centers in the United States. Ann Intern Med. 2002 Dec 17;137(12):947-54. doi: 10.7326/0003-4819-137-12-200212170-00007. PMID 12484709
- [Background] Fountain FF, Tolley E, Chrisman CR, Self TH. Isoniazid hepatotoxicity associated with treatment of latent tuberculosis infection: a 7-year evaluation from a public health tuberculosis clinic. Chest. 2005 Jul;128(1):116-23. doi: 10.1378/chest.128.1.116. PMID 16002924
- [Background] Kopanoff DE, Snider DE Jr, Caras GJ. Isoniazid-related hepatitis: a U.S. Public Health Service cooperative surveillance study. Am Rev Respir Dis. 1978 Jun;117(6):991-1001. doi: 10.1164/arrd.1978.117.6.991. PMID 666111
- [Background] International Union Against Tuberculosis Committee on Prophylaxis. Efficacy of various durations of isoniazid preventive therapy for tuberculosis: five years of follow-up in the IUAT trial. International Union Against Tuberculosis Committee on Prophylaxis. Bull World Health Organ. 1982;60(4):555-64. PMID 6754120
- [Background] Steele MA, Burk RF, DesPrez RM. Toxic hepatitis with isoniazid and rifampin. A meta-analysis. Chest. 1991 Feb;99(2):465-71. doi: 10.1378/chest.99.2.465. No abstract available. PMID 1824929
- [Background] Thongraung W, Sittidach M, Khwansuwan P, Sariyasuntorn K, Wongsampan S. Evaluation of the physicians' approach to the diagnosis and treatment of patients with antituberculosis drug-induced hepatotoxicity. J Eval Clin Pract. 2012 Dec;18(6):1119-25. doi: 10.1111/j.1365-2753.2011.01706.x. Epub 2011 Jun 22. PMID 21696520
- [Background] Huang YS, Chern HD, Su WJ, Wu JC, Lai SL, Yang SY, Chang FY, Lee SD. Polymorphism of the N-acetyltransferase 2 gene as a susceptibility risk factor for antituberculosis drug-induced hepatitis. Hepatology. 2002 Apr;35(4):883-9. doi: 10.1053/jhep.2002.32102. PMID 11915035
- [Background] Yang S, Hwang SJ, Park JY, Chung EK, Lee JI. Association of genetic polymorphisms of CYP2E1, NAT2, GST and SLCO1B1 with the risk of anti-tuberculosis drug-induced liver injury: a systematic review and meta-analysis. BMJ Open. 2019 Aug 1;9(8):e027940. doi: 10.1136/bmjopen-2018-027940. PMID 31375612